CLINICAL TRIAL: NCT04933565
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Bioavailability of ORG-129 After Single and Multiple Ascending Oral Doses (Including Food Interaction Effect) in Healthy Young Volunteers
Brief Title: First in Human Study of ORG-129 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Origo Biopharma (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ORG129-CT01
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORG-129 (Experimental): Single ascending dose (up to 4 cohorts), Multiple ascending dose (up to 4 cohorts), Food interaction cohort, Multiple dose PK/PD cohort
  Interventions: Drug: ORG-129
- Placebo (Placebo Comparator): Single ascending dose (up to 4 cohorts), Multiple ascending dose (up to 4 cohorts), Food interaction cohort, Multiple dose PK/PD cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORG-129 — ORG-129 oral capsules
  Arms: ORG-129
Drug: Placebo — Placebo oral capsules
  Arms: Placebo

SUMMARY:
The current study is performed to characterize the safety, tolerability and pharmacokinetics of ORG-129 after oral intake in healthy male and female volunteers after single ascending and multiple ascending doses.

ELIGIBILITY:
Inclusion Criteria:

To be included in the Single Dose Study, subjects should meet all the following criteria at the screening visit:

1. Healthy male subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination.
4. Laboratory tests (hematology and biochemistry) within the range of normal values, according to the Biochemistry laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50- 100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
7. To be able to understand the nature of the study and comply with all their requirements.
8. Free acceptance to participate in the study should be stated in an informed consent document signed by the volunteer which must be approved by the CREC.

For the Multiple Dose Study, subjects should meet all the following inclusion criteria at screening visit:

1. Healthy male/female subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination at screening and baseline.
4. Laboratory tests (hematology, biochemistry and urianalysis) within the range of normal values, according to the laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50- 100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
7. Females must be of non-childbearing potential (i.e., surgically sterile) or have to use contraceptive measures (non-hormonal) such as condom, diaphragm or cervical/vault cap with spermicide until 28 days post-administration.
8. To be able to understand the nature of the study and comply with all their requirements.
9. Free acceptance to participate in the study by obtains signed informed consent form approved by the CREC.

Exclusion Criteria:

For the single dose study and multiple dose study meeting any of the following criteria at screening visit will be excluded from entry into the study:

1. History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 gr/day for men and >24 for women (in MAD).
2. Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day) and grape juice.
3. Background of idiosyncrasy, food intolerance, hypersensitivity or adverse reactions to any drug or galenical form.
4. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
5. Intake of any medication within 2 weeks prior taking the study treatment (except for use of paracetamol in short-term symptomatic treatments), including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), or any enzymatic inductor or inhibitor within 3 months before the drug administration.
6. Positive serology for hepatitis B, C or HIV.
7. Background or clinically significant evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological disease or other chronic diseases.
8. History of psychiatric diseases or epileptic seizures.
9. 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
10. Having undergone major surgery during the previous 6 months.
11. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc.) from 6 months prior to drug administration.
12. Participation in other clinical trials during the previous 90 days (last drug to first drug administration period) in which an investigational drug or a commercially available drug was tested.
13. Donation of blood during the 4 weeks preceding the drug administration.
14. Severe or moderate acute illness 4 weeks before drug administration.
15. Clinically significant infections within 3 months or any infection within 28 days of screening.
16. History or recurrent disseminated herpes simplex or herpes zoster.
17. Personal or family history of hereditary immunodeficiency
18. Clinically significant abnormal laboratory values (as determined by the PI) at the screening evaluation.
19. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract
20. Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the PI).
21. Females with positive results from the pregnancy test or breast-feeding (MAD).
22. Females with hormonal contraceptive therapy.
23. Positive Covid-19 diagnosis prior to hospital admission

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SAD of ORG-129 | day 1 through day 8
  by assessing the number, severity and type of treatment emergent adverse events
To assess the safety and tolerability of MAD of ORG-129 | day 1 through day 12
  by assessing the number, severity and type of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics of ORG-129 when given as SAD: AUC | Day 1 and Day 2
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics of ORG-129 when given as SAD: Cmax | Day 1 and Day 2
  Maximum observed concentration (Cmax)
Pharmacokinetics of ORG-129 when given as SAD: Tmax | Day 1 and Day 2
  Time to reach maximum observed concentration (Tmax)
Pharmacokinetics of ORG-129 when given as SAD: CL/F | Day 1 and Day 2
  Oral Clearance (CL/F)
Pharmacokinetics of ORG-129 when given as SAD: Vz/F | Day 1 and Day 2
  Terminal Phase Volume of Distribution(Vz/F)
Pharmacokinetics of ORG-129 when given as SAD: Kel | Day 1 and Day 2
  Elimination Rate (Kel)
Pharmacokinetics of ORG-129 when given as SAD: t 1/2 | Day 1 and Day 2
  Elimination Halflife (t 1/2)
Pharmacokinetics of ORG-129 when given as MAD: AUC | Day 1 and Day 5
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics of ORG-129 when given as MD: AUC | Day 1 and Day 10
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics of ORG-129 when given as MAD: Cmax | Day 1 and Day 5
  Maximum observed concentration (Cmax)
Pharmacokinetics of ORG-129 when given as MD: Cmax | Day 1 and Day 10
  Maximum observed concentration (Cmax)
Pharmacokinetics of ORG-129 when given as MAD: Tmax | Day 1 and Day 5
  Time to reach maximum observed concentration (Tmax)
Pharmacokinetics of ORG-129 when given as MD: Tmax | Day 1 and Day 10
  Time to reach maximum observed concentration (Tmax)
Pharmacokinetics of ORG-129 when given as MAD: CL/F | Day 1 and Day 5
  Oral Clearance (CL/F)
Pharmacokinetics of ORG-129 when given as MD: CL/F | Day 1 and Day 10
  Oral Clearance (CL/F)
Pharmacokinetics of ORG-129 when given as MAD: Vz/F | Day 1 and Day 5
  Terminal Phase Volume of Distribution(Vz/F)
Pharmacokinetics of ORG-129 when given as MD: Vz/F | Day 1 and Day 10
  Terminal Phase Volume of Distribution(Vz/F)
Pharmacokinetics of ORG-129 when given as MAD: Kel | Day 1 and Day 5
  Elimination Rate (Kel)
Pharmacokinetics of ORG-129 when given as MD: Kel | Day 1 and Day 10
  Elimination Rate (Kel)
Pharmacokinetics of ORG-129 when given as MAD: t 1/2 | Day 1 and Day 5
  Elimination Halflife (t 1/2)
Pharmacokinetics of ORG-129 when given as MD: t 1/2 | Day 1 and Day 10
  Elimination Halflife (t 1/2)
Pharmacokinetics of ORG-129 when given as MAD: Css | Day 5
  concentration at steady state (Css)
Pharmacokinetics of ORG-129 when given as MD: Css | Day 10
  concentration at steady state (Css)
PK of ORG-129 when given as MAD: C trough [ Time Frame: Day 2, 5 ] | Day 2 and Day 5
  C trough
PK of ORG-129 when given as MD: C trough [ Time Frame: Day 2, 10 ] | Day 2 and Day 10
  C trough
PD of ORG-129 when given as MD [ Time Frame: Day 2, 10 ] | Day 1-10
  Biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: Juan Martinez-Colomer, MD, Principal Investigator — Institut de Recerca de l'Hospital de la Santa Creu i de Sant Pau
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i de Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No